CLINICAL TRIAL: NCT02328781
Title: Prospective Multi-center Single-arm Target Value Clinical Trial for Evaluating Clinical Use Safety and Efficacy of the Firehorus Vertebral Artery Rapamycin-target-eluting Stent System
Brief Title: Prospective Evaluation of Safety and Efficacy Vertebral Drug-eluting Stent System
Acronym: PESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongrong Miao (Other)
Responsible Party: Sponsor-Investigator, Zhongrong Miao, Chief of Interventional Neuroloy Department, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTH-PESS; NCT03859674 (obsolete NCT alias)
Record Dates: First submitted 2014-12-28; First posted 2014-12-31 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Vertebrobasilar Insufficiency
Keywords: vertebral artery stenosis; drug-eluting stent
MeSH Terms: conditions — Vertebrobasilar Insufficiency | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Drug-eluting stent
  Interventions: Device: Drug-eluting stent

INTERVENTIONS:
Device: Drug-eluting stent

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Firehorus vertebral artery rapamycin-target-eluting stent system (hereinafter referred to as Firehorus) in treatment of symptomatic vertebral artery stenosis.

DETAILED DESCRIPTION:
This clinical trial utilizes the prospective, multicenter, single-arm target value trial design, to evaluate the safety and efficacy of Firehorus vertebral artery rapamycin-target-eluting stent system (hereinafter referred to as Firehorus) in clinical use, for which 5 (or more) institutions will be selected as Clinical Trial Centre.Subjects will be screened in accordance with the inclusion and exclusion criteria of the this protocol and will be treated with Firehorus. Immediate stent implantation success rate of all subjects after surgery will be recorded, DSA angiographic follow-up will be performed at six months (±30 days) after surgery to assess the incidence of stent restenosis ( stenosis ≥ 50%) of the subjects, and the subjects will be followed up at 30 days (±7 days), 6 months (± 30 days), 12 months (± 30 days) after surgery , so as to evaluate the safety and efficacy of Firehorus in clinical use. The expected participating duration of each subject from enrollment to complete the follow-up is 12 months (± 30 days).

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years (including 18 years old), and under 80 years old (including 80 years old), male / Pregnancy Test ( -) female
2. Patients with symptomatic vertebral artery stenosis not responding to drug therapy (defined as stroke or TIA occurred within 90 days, the patient is using at least one antithrombotic drug and receiving interventions for other vascular risk factors, such as antihypertensive therapy or lipid-lowering therapy for hypertensionor high cholesterol when stroke or TIA occurs)
3. DSA angiography indicated target lesion stenosis ≥ 50% (the degree of stenosis is determined according to the WASID method)
4. Length of vascular lesion ≤ 21mm
5. Modified Rankin score < 3
6. Suiform for placing with vertebral artery rapamycin-eluting stent, voluntary to receive follow-up and sing the informed consent

Exclusion Criteria:

1. There is a series of stenosis lesion within the target lesion region
2. TIA or non- disabling stroke (such as atrial fibrillation, etc.) caused by other factors other than vertebral artery stenosis
3. The target lesion area had received previous surgery or endovascular treatment
4. Combined with severe systemic disease or with other disease with the potential risk to cause fatal sudden illness, or the subject with life expectancy <2 years
5. Unsuitable / intolerable to dual antiplatelet therapy
6. Suffered from cerebral infarction and severe neurological dysfunction related to the responsible blood vessels (modified Rankin score ≥ 3 points)
7. Experienced severe myocardial infarction within 2 weeks
8. Accompanied by other intracranial lesions, such as intracranial hemorrhage, aneurysm, arteriovenous malformations, brain tumors, etc.
9. Arterial dissection, moyamoya disease, arteritis active, unexplained non- atherosclerotic stenosis
10. Serious target vessel tortuosity / calcification, leading to not suitable for stenting / lesion can not be expanded
11. Severe renal impairment, or allergic to or resistant to contrast agent, rapamycin (Rapamycin) and its derivatives, cobalt based alloys, polylactic acid ;
12. Patients participated in other drugs or equipment and have not reached the endpoint
13. The patient or their family members do not agree to sign an informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
rate of in-stent restenosis | 6 months (± 30 days) after procedure
  DSA angiography performed after 6 months (± 30 days) showed the occurrence of in-stent restenosis and the restenosis rate ≥ 50%;

SECONDARY OUTCOMES:
Immediate stent implantation success rate | Immediate after the procedure
  postoperative angiography immediately after implantation of Firehorus indicated that residual stenosis ≤ 20% (the degree of stenosis is determined according to the WASID method)
Any death or stroke related to the treated area | 1 year
  Any death or stroke related to the treated area supplied by the target blood vessels during the follow-up period.
Any death or stroke | 1 year
  Any death or stroke during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, PhD,MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China